CLINICAL TRIAL: NCT01472952
Title: System-level Monitoring of Immune Activation Concerning Susceptibility to Sepsis in Trauma Patients
Status: Withdrawn | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Timo Sturm, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2011-211N-MA
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Trauma; Sepsis
Keywords: sepsis; immune cells; immune reaction; trauma; Immune activation
MeSH Terms: conditions — Wounds and Injuries; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sepsis remains a common entity in critical care patients with remarkable mortality. Despite extended research activities, no reliable bio-markers or scoring systems attributing the individual risk of developing sepsis have been found so far.

Patients with multiple trauma are at high risk of developing sepsis. Due to local and systemic immune reactions, high plasma levels of known pro-inflammatory cytokines can be found.

Simultaneously, certain anti-inflammatory reactions such as changes in immune cell activity and serum cytokine levels, known as "compensatory anti-inflammatory response syndrome" (CARS) take place.

In addition to changes of cytokine levels and immune cell activity, underlying genetic reactions are present. For instance, expression of miRNA (as an potential important step of immune cell activation) is likely changed during systemic and local immune reactions.

In the present study levels of pro- and antiinflammatory cytokines, a detailed assay of immune cell activation and the various expression of miRNA will be evaluated in patients of multiple trauma on day 1 and day 4.

Additionally, clinical parameters of organ function, current infection markers as CRP and Procalcitonin, cardiovascular function such as Indocyanin clearance and hemodynamic measures delivered with PiCCO-system and heart rate variability will be assessed. Parameters of local tissue perfusion will be measured with transcutaneous laser doppler.

ELIGIBILITY:
Inclusion Criteria:

* multiple trauma,
* ISS > 16

Exclusion Criteria:

* resuscitation
* pregnancy
* malignancy
* chronic renal insufficiency
* steroid intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critical care patients with multiple trauma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Sepsis | 14 days